CLINICAL TRIAL: NCT06361602
Title: Exploring the Effectiveness and Factors Affecting the Collection of Single Nucleated Cells From Different Volunteers
Acronym: SYX-AN-01
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-1015-01
Record Dates: First submitted 2024-03-26; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Observational Study

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: inapplicable — inapplicable

SUMMARY:
1. 80 cases of healthy donors were subjected to peripheral blood single nucleated cells (PBMC) collection and analyzed the effects of age, body mass index (BMI), blood routine indexes before collection, collection of circulating blood volume, volume of processed blood and the number of circulations, etc., on the PBMC obtained from both men and women, and explored the effects of PBMC collection in different volunteers and the factors affecting the collection. and the influencing factors.
2. The data obtained will provide a reference for the MNC threshold for the subsequent clinical trials of immunocell therapy in hospitals.
3. From the screening of volunteers, PBMC collection and transportation conditions and other specific details of the operation, risk assessment and the establishment of a safe operation standard process, for the hospital to carry out subsequent clinical trials of immune cell therapy to provide an effective reference.

DETAILED DESCRIPTION:
1. Nationality is not limited, age is 18-55 years old (including boundary value), gender is not limited;
2. Body weight: male ≥ 50kg, female ≥ 45kg and 18.5kg/m2 ≤ BMI ≤ 30kg/m2 (BMI, body mass index = weight (kg) ÷ height (m)2);
3. Blood pressure:

   12.0Kpa (90mmHg)≤systolic blood pressure≤18.7Kpa (140mmHg) 8.0Kpa (60mmHg) ≤ diastolic blood pressure ≤ 12.0Kpa (90mmHg);
4. Pulse: 60 beats/min ≤ pulse ≤ 100 beats/min, ≥ 50 beats/min for high endurance athletes, or rhythmic abnormalities without clinical significance;
5. Ear temperature: 35.7 ≤ body temperature ≤ 37.5 ℃;
6. Good general condition of the body: no damage to vital organs such as heart, lungs, liver, kidneys, etc., no serious or uncontrolled infections, no history of serious mental disorders;
7. Clinical examination should fulfill the following criteria:

7.1 Hemoglobin (Hb) measurement is normal or abnormal without clinical significance; 7.2 White blood cell (WBC) measurement: (3.5-10) × 109/L; 7.3 Platelet count (PLT) determination normal or abnormal without clinical significance; 7.4 Neutrophil count (NEU) determination normal or abnormal without clinical significance; 7.5 Normal or abnormal liver and kidney function test indexes without clinical significance; 7.6 Normal or abnormal coagulation function without clinical significance; 7.7 Hepatitis B virus surface antigen (HBsAg) negative; 7.8 Hepatitis C virus antibody (HCV antibody) negative; 7.9 human immunodeficiency virus antibody (HIV-1 and HIV-2 antibody) negative; 7.10 Syphilis negative;

ELIGIBILITY:
Inclusion Criteria.

1. No restriction on nationality, age 18-55 years old (including borderline value), no restriction on gender;
2. Body weight: Male ≥50kg, female ≥45kg and 18.5kg/m2≤BMI≤30kg/m2 (BMI=Body Mass Index (BMI) = Weight (kg)÷Height (m)2);
3. Blood pressure:

   12.0Kpa (90mmHg)≤systolic blood pressure≤18.7Kpa (140mmHg) 8.0Kpa (60mmHg) ≤ diastolic blood pressure ≤ 12.0Kpa (90mmHg);
4. Pulse: 60 beats/min ≤ pulse ≤ 100 beats/min, ≥ 50 beats/min for high endurance athletes, or rhythmic abnormalities without clinical significance;
5. Ear temperature: 35.7 ≤ body temperature ≤ 37.5 ℃;
6. Good general condition of the body: no damage to vital organs such as heart, lungs, liver, kidneys, etc., no serious or uncontrolled infections, no history of serious mental disorders;
7. Clinical examination should fulfill the following criteria:

7.1 Hemoglobin (Hb) measurement is normal or abnormal without clinical significance; 7.2 White blood cell (WBC) measurement: (3.5-10) × 109/L; 7.3 Platelet count (PLT) determination normal or abnormal without clinical significance; 7.4 Neutrophil count (NEU) determination normal or abnormal without clinical significance; 7.5 Normal or abnormal liver and kidney function test indexes without clinical significance; 7.6 Normal or abnormal coagulation function without clinical significance; 7.7 Hepatitis B virus surface antigen (HBsAg) negative; 7.8 Hepatitis C virus antibody (HCV antibody) negative; 7.9 human immunodeficiency virus antibody (HIV-1 and HIV-2 antibody) negative; 7.10 Syphilis negative;

Exclusion Criteria.

1. the following diseases considered clinically significant by the investigator: 1.1 Have respiratory, circulatory, gastrointestinal, urinary, hematologic, immunologic, endocrine system diseases or metabolic disorders; neurological disorders, psychiatric disorders, Creutzfeldt-Jakob disease, and those with a family history of the disease, or those who are receiving treatment with tissues or tissue derivatives that may have originated from infection with Creutzfeldt-Jakob pathogens; 1.2 Persons with chronic skin diseases, especially infectious, allergic or inflammatory systemic skin diseases; persons with allergic diseases or recurrent allergic attacks; 1.3 persons with malignant tumors or benign tumors affecting health;
2. those who have not completed 3 months of minor surgery, such as appendectomy, ophthalmic surgery after healing, etc.; those who have not completed 1 year of major surgery, such as: benign gynecological tumors, gastrointestinal malignant tumors after surgery, etc;
3. Women during pregnancy, less than 6 months after abortion, and less than 1 year after delivery and breastfeeding;
4. Less than 1 week after recovering from upper respiratory tract infection or less than 3 months after recovering from pneumonia;
5. less than 3 months after recovery from acute pyelonephritis, or during the period of urinary stone attack;
6. Injury caused by equipment contaminated by blood or tissue fluid or contaminated wounds, or less than 1 year after tattooing;
7. Those who have received whole blood and blood component transfusion within 1 year;
8. within 2 weeks after the last vaccination with live attenuated measles, mumps, or polio vaccine, or within 4 weeks after the last immunization with live rubella vaccine or live attenuated encephalitis B vaccine;
9. Within 1 year after the last immunization with rabies vaccine after being bitten by an animal;
10. within 4 weeks of the last immunization with antitoxin or immune serum injection or within 1 year of the last immunization with hepatitis B human immunoglobulin injection
11. those who have a documented clinical trial with leukocyte, plasma, platelet, or whole blood donation within 3 months
12. who, in the opinion of the investigator, are not suitable for participation in this study.

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Healthy volunteers of any nationality, aged 18-55 (including boundary values) and of any gender
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Exploring the effectiveness and factors affecting the collection of single nucleated cells from different volunteers | MAY 1, 2027
  We collected peripheral blood single nucleated cells (PBMC) from 80 healthy donors and analyzed the effects of age, body mass index (BMI), pre-collection blood parameters, collection of circulating blood volume, volume of processed blood, and the number of circulations on the PBMC collected from both male and female donors, to explore the effects of different volunteers on the collection of PBMC and the factors affecting the collection of PBMC. The effect of PBMC collection in different volunteers and the influencing factors were investigated.